CLINICAL TRIAL: NCT07009860
Title: RESTORE TRIAL: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Pemvidutide in the Treatment of Alcohol-Associated Liver Disease (ALD)
Brief Title: RESTORE TRIAL: A Phase 2 Study Evaluating the Efficacy and Safety of Pemvidutide in the Treatment of Alcohol-Associated Liver Disease (ALD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-801-241
Record Dates: First submitted 2025-06-05; First posted 2025-06-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pemvidutide 2.4 mg (Experimental)
  Interventions: Drug: Pemvidutide
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pemvidutide — Pemvidutide 2.4 mg
  Arms: Pemvidutide 2.4 mg
Other: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of pemvidutide in subjects with ALD.

* Pemvidutide: 2.4 mg SC once weekly
* Placebo: Placebo SC once weekly

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 18 to 75 years, inclusive
2. Overweight or obesity, defined as BMI ≥ 25 kg/m2
3. History of alcohol misuse for the prior 3 years, with an alcohol intake ≥ 50 grams per day for males and ≥ 40 grams per day for females on average in the past year
4. Liver stiffness of 10.0-18.5 kPa by VCTE, inclusive

Exclusion Criteria:

1. Presence of clinically significant alcohol withdrawal symptoms, defined as CIWA-Ar score ≥ 10 at screening and/or prior to randomization
2. History of hospitalization for alcohol intoxication or alcohol withdrawal within the past year
3. History of seizures related to alcohol within the past year
4. History and/or current DSM-5 diagnosis of schizophrenia, bipolar disorder, psychotic disorder, or another severe psychiatric disorder, unless documented as well-controlled by the Investigator for at least 6 months prior to screening and cleared by the Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Relative (%) change in liver stiffness by VCTE compared to baseline at Week 24 | Week 24

SECONDARY OUTCOMES:
Relative (%) change in liver stiffness by VCTE compared to baseline at Week 48 | Week 24 and 48
Absolute change in the Enhanced Liver Fibrosis (ELF) score at Weeks 24 and 48 compared to baseline | Week 24 and 48

CONTACTS AND LOCATIONS:
Locations (33):
- United States (32):
  - Altimmune Clinical Study Site, Peoria, Arizona
  - Altimmune Clinical Study Site, Tucson, Arizona
  - Altimmune Clinical Study Site, North Little Rock, Arkansas
  - Altimmune Clinical Study Site, Fresno, California
  - Altimmune Clinical Study Site, La Jolla, California
  - Altimmune Clinical Study Site, Pasadena, California
  - Altimmune Clinical Study Site, Englewood, Colorado
  - Altimmune Clinical Study Site, Bradenton, Florida
  - Altimmune Clinical Study Site, Doral, Florida
  - Altimmune Clinical Study Site, Fort Myers, Florida
  - Altimmune Clinical Study Site, Miami, Florida
  - Altimmune Clinical Study Site, Miami Lakes, Florida
  - Altimmune Clinical Study Site, Naples, Florida
  - Altimmune Clinical Study Site, Orlando, Florida
  - Altimmune Clinical Study Site, Port Orange, Florida
  - Altimmune Clinical Study Site, Atlanta, Georgia
  - Altimmune Clinical Study Site, Indianapolis, Indiana
  - Altimmune Clinical Study Site, Louisville, Kentucky
  - Altimmune Clinical Study Site, Bastrop, Louisiana
  - Altimmune Clinical Study Site, Marrero, Louisiana
  - Altimmune Clinical Study Site, Kansas City, Missouri
  - Altimmune Clinical Study Site, Las Vegas, Nevada
  - Altimmune Clinical Study Site, Manhasset, New York
  - Altimmune Clinical Study Site, Westlake, Ohio
  - Altimmune Clinical Study Site, Brownsville, Texas
  - Altimmune Clinical Study Site, Dallas, Texas
  - Altimmune Clinical Study Site, Edinburg, Texas
  - Altimmune Clinical Study Site, Houston, Texas
  - Altimmune Clinical Study Site, San Antonio, Texas
  - Altimmune Clinical Study Site, Waco, Texas
  - Altimmune Clinical Study Site, Richmond, Virginia
  - Altimmune Clinical Study Site, Seattle, Washington
- Altimmune Clinical Study Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that the results of this study will be presented at scientific meetings and/or published in a peer reviewed scientific or medical journal. A Publications Committee, comprised of the Investigators participating in the study and representatives from the Sponsor, as appropriate, will be formed to oversee the publication of the study results, which will reflect the experience of all participating study centers. Subsequently, individual Investigators may publish results from the study in compliance with their agreement with the Sponsor.